CLINICAL TRIAL: NCT02491203
Title: Maximizing Post-stroke Upper Limb Rehabilitation Using a Novel Telerehabilitation Interactive Virtual Reality System in the Patient's Home
Brief Title: Post-stroke Upper Limb Rehabilitation Using Telerehabilitation Interactive Virtual Reality System in the Patient's Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Dahlia Kairy, Professor, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRIR-937-0214
Record Dates: First submitted 2015-06-13; First posted 2015-07-07 (Estimated); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Stroke
Keywords: Virtual reality; telerehabilitation; Stroke rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention): All study participants in the control group will receive a 4-week written home exercise program (e.g. GRASP) , i.e. the usual care discharge home program.
- Telerehabilitation system (Experimental): Participants in the experimental group will receive four weeks written home exercise program provided by a clinician, i.e. usual care discharge home program plus virtual reality (VR) and telerehabilitation system. The intensity and choice of game for the home program will be determined by the therapist based on the patient's abilities, interests, motivation and fatigue. The patient's performance for the VR home program will be monitored asynchronously and the program adapted to ensure it remains at an appropriate level for the patient.
  Interventions: Other: Telerehabilitation system

INTERVENTIONS:
Other: Telerehabilitation system — Usual care plus home-based virtual reality telerehabilitation system.
  Arms: Telerehabilitation system

SUMMARY:
Stroke is a leading cause of death and long-term disability worldwide and its incidence is on the rise. Importantly, loss of arm function occurs in up to 85% of stroke survivors, with a significant long-term impact on activities of daily living, leisure activities and work. The capacity for recovery following a stroke depends on several factors, including the extent of the initial neurological damage, spontaneous recovery and rehabilitation, with possible recovery even years after the stroke. Unfortunately, accessibility of much needed rehabilitation services poststroke often remains limited, both in terms of intensity and duration, as reported in a recent report on post-stroke rehabilitation services in Quebec (Richard, 2013) Recent evidence suggests that homebased telerehabilitation (TR) is a viable approach for upper limb training post-stroke when rehabilitation services are not available. Similarly, the Canadian Best Practice Recommendations for Stroke Care update for 2013 recommends home-based patient monitoring be used when frequent monitoring is needed and face-to-face visits are not available. Hence, The investigators have developed and propose to examine the use of a TR system that allows upper limb rehabilitation with ongoing off-line monitoring, to be used after usual poststroke rehabilitation is completed and services are no longer offered.

DETAILED DESCRIPTION:
More specifically, the objective of the proposed study is to assess the impact, in terms of motor recovery, function,quality of life, compliance, safety and cost, of a novel, patient-centered home-based tailored TR program using an affordable virtual reality system for upper-limb rehabilitation post-stroke. Such a system, combined with remote off-line monitoring could allow patients to take charge and pursue their rehabilitation beyond current services, maximizing their potential for recovery.

A single-blind two-arm randomized clinical trial (RCT) is proposed for this study with participants who have had a stroke randomly allocated to: (1) 4-week training with home-based tele-rehabilitation (TR) system (see intervention below).i.e. treatment group or (2) 4-week written home exercise program provided by a clinician, i.e. exercise control group.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or hemorrhagic stroke (does not have to be a first time stroke);
* Mild to moderate upper limb impairment (score 3-6 Chedoke-McMaster arm component or ability to perform VR tasks at least at the lowest setting according to clinician);
* At least 6 months post stroke;
* No longer receiving rehabilitation services; and (5) living in an area where high speed Internet access is available.

Exclusion Criteria:

* Being medically unstable;
* Severe cognitive or communication deficits;
* Visual impairments;
* Severe balance deficits limiting sitting safely independently;
* Shoulder pain;
* Previous upper limb impairment limiting potential recovery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-09; Primary Completion 2016-09 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Upper limb motor control at 4 weeks | baseline and four weeks after intervention
  as measured using the Fugl-Meyer Assessment-UE (FMA-UE).

SECONDARY OUTCOMES:
Change from Baseline in quality of life at 4 weeks | At intake into the study ( post-stroke; chronic phase) and four weeks after intervention
  measured using the Stroke Impact Scale-16, a stroke-specific, self-report, health status measure featuring 16 items capturing daily activities
Change from Baseline in Upper limb motor control at 4 weeks | At intake into the study ( post-stroke; chronic phase) and four weeks after intervention
  Box and Block test.
Change from Baseline in Upper limb function at 4 weeks | At intake into the study ( post-stroke; chronic phase) and four weeks after intervention
  Impact on upper extremity use in daily activities will be using the Motor Activity Log, a self-reported measure of upper limb use

OTHER OUTCOMES:
Economic evaluation at 4 weeks after intervention | at 4 weeks after intervention
  Cost-effectiveness analysis (CEA) comparing the intervention with usual care

CONTACTS AND LOCATIONS:
Overall Officials: Dahlia Kairy, PhD, Principal Investigator — Université de Montréal
Locations (1):
- University of Montreal, Montreal, Quebec, Canada

REFERENCES:
- [Background] Feigin VL, Lawes CM, Bennett DA, Barker-Collo SL, Parag V. Worldwide stroke incidence and early case fatality reported in 56 population-based studies: a systematic review. Lancet Neurol. 2009 Apr;8(4):355-69. doi: 10.1016/S1474-4422(09)70025-0. Epub 2009 Feb 21. PMID 19233729
- [Background] Roger VL, Go AS, Lloyd-Jones DM, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Soliman EZ, Sorlie PD, Sotoodehnia N, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2012 update: a report from the American Heart Association. Circulation. 2012 Jan 3;125(1):e2-e220. doi: 10.1161/CIR.0b013e31823ac046. Epub 2011 Dec 15. No abstract available. PMID 22179539
- [Background] Nichols-Larsen DS, Clark PC, Zeringue A, Greenspan A, Blanton S. Factors influencing stroke survivors' quality of life during subacute recovery. Stroke. 2005 Jul;36(7):1480-4. doi: 10.1161/01.STR.0000170706.13595.4f. Epub 2005 Jun 9. PMID 15947263
- [Background] Richards C. Trajectoires de services de réadaptation post-AVC. Un continuum centré sur la personne: Comité d'experts sur l'offre de services de réadaptation post-AVC;2013
- [Background] Langan J, Delave K, Phillips L, Pangilinan P, Brown SH. Home-based telerehabilitation shows improved upper limb function in adults with chronic stroke: a pilot study. J Rehabil Med. 2013 Feb;45(2):217-20. doi: 10.2340/16501977-1115. PMID 23319181
- [Background] Dawson AS KJ MA, Foley N, Teasell R. Chapter 5: Stroke Rehabilitation. In: Lindsay MP GG BM, Phillips S, ed. Canadian Best Practice Recommendations for Stroke Care: Canadian Stroke Best Practices and Standards Working Group; 2013.
- [Derived] Hernandez A, Bubyr L, Archambault PS, Higgins J, Levin MF, Kairy D. Virtual Reality-Based Rehabilitation as a Feasible and Engaging Tool for the Management of Chronic Poststroke Upper-Extremity Function Recovery: Randomized Controlled Trial. JMIR Serious Games. 2022 Sep 27;10(3):e37506. doi: 10.2196/37506. PMID 36166289